CLINICAL TRIAL: NCT06142396
Title: Pilot Study of Daratumumab in Combination With Bortezomib, Cyclophosphamide, and Dexamethasone (Dara-CyBorD) in Newly Diagnosed Multiple Myeloma Patients With Renal Failure
Brief Title: Pilot Study Dara-CyBorD in Newly Diagnosed Multiple Myeloma Patients With Renal Failure
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54767414MMY2095
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Renal Failure
Keywords: Daratumumab; Bortezomib; Cyclophosphamide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Pilot study for combination medication treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dara-CyBorD (Experimental): Induction treatment with daratumumab-hyaluronidase (dara SC) in combination with cyclophosphamide, bortezomib, and dexamethasone (Dara-CyBorD) for four cycles of 28 days, followed by restaging with repeat PET-CT, bone marrow evaluation, and myeloma serological testing.
  Interventions: Combination Product: Daratumumab-hyaluronidase in Combination with Bortezomib, Cyclophosphamide, and Dexamethasone

INTERVENTIONS:
Combination Product: Daratumumab-hyaluronidase in Combination with Bortezomib, Cyclophosphamide, and Dexamethasone — This intervention is Daratumumab-hyaluronidase in combination with the chemotherapy regimen "CyBord" (cyclophosphamide, bortezomib, and dexamethasone) and then with lenalidomide maintenance in patients with newly diagnosed multiple myeloma who have new onset renal failure.
  Other Names: DaraCyBord

SUMMARY:
The goal of this study is to assess the efficacy of induction treatment with daratumumab-hyaluronidase (dara SC) with cyclophosphamide, bortezomib, and dexamethasone (Dara-CyBorD) for four cycles in patients with newly diagnosed multiple myeloma who have new onset renal failure. This study will also investigate the difference responses in African American (AA) patients versus non-African American patients.

The primary questions this study aims to answer are:

1. To evaluate the very good partial response rate (VGPR) after 4 cycles of Dara-CyBord.
2. To evaluate the renal response rate (RRR) after 4 cycles of Dara-CyBord.

DETAILED DESCRIPTION:
Acute renal impairment (RI) is a myeloma emergency. Diagnosis should be established as fast as possible, and antimyeloma therapy should be started immediately after confirmation of the diagnosis to restore renal function rapidly. The incidence of RI at diagnosis ranges from 20% to 50%. Patients with RI had more advanced disease than the others, a lower response rate to treatment than those with normal renal function, and shorter survival. Overall survival is significantly longer among those with baseline CrCl ≥30 mL per minute than those with CrCl <30 mL per minute.

This is a prospective, interventional pilot study for patients with newly diagnosed multiple myeloma (NDMM) who have new onset renal failure. The study will implement a planned enrollment strategy to focus on the African American (AA) patient population, with an accrual goal of 50% of all participants. All participants will be assigned to receive induction treatment with daratumumab-hyaluronidase (dara SC) with cyclophosphamide, bortezomib, and dexamethasone (Dara-CyBorD) for four cycles of 28 days, followed by restaging with repeat PET-CT, bone marrow evaluation, and myeloma serological testing. After induction with Dara-CyBorD, further treatment as per standard guidelines will be determined at the physician's discretion based on transplant eligibility to either an additional 2 cycles of Dara-CyBorD followed by maintenance therapy (if transplant ineligible) or autologous stem cell transplantation (ASCT) followed by maintenance therapy (if transplant eligible). Maintenance therapy will consist of lenalidomide with dara SC for 2 years. Participants will be followed every three months for up to 2 years per the standard guidelines or until disease progression or the start of a new line of therapy to assess the duration of response.

The use of novel antimyeloma agents resulted in a substantial increase in the survival of patients with MM with RI. MM patients with RI are generally excluded from clinical trials. Clinical trials for MM patients with RI are an unmet need. Bortezomib-based regimens remain the cornerstone of the management of myeloma-related RI, with high-dose dexamethasone, with the addition of a conventional chemotherapy agent (cyclophosphamide).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have had a confirmed new diagnosis of MM following revised IMWG criteria.
2. Patients must have Zubrod/ECOG Performance Status ≤ 2.
3. Patients must have renal insufficiency. Renal insufficiency is defined as eCrCl < 60 mL/min (using Cockcroft-Gault Equation for Cr Cl) and/or necessitating dialysis
4. must not have known allergies to any of the study drugs. Must have adequate organ function.
5. International normalized ratio (INR) and prothrombin time (PT) ≤1.5 × ULN. Activated partial thromboplastin time (aPTT) ≤1.5 × ULN.

Exclusion Criteria:

* 1. Known seropositive for: human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.

  2. Known Chronic obstructive pulmonary disease (COPD). 3. Known Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification.

  4. Known Clinically significant heart disease is defined as: myocardial infarction within 6 months before enrollment, or unstable or uncontrolled disease/condition related to or affection cardiac function.

  5. Women who are pregnant, breastfeeding, or planning to become pregnant while enrolled in this study.

  6. Patients with grade 3 or 4 peripheral neuropathy 7. Patients with other active malignancies that require concurrent treatment 8. Known CNS involvement or plasma cell leukemia, or AL amyloidosis 9. Participants with active infection requiring systemic therapy 10. Has known substance abuse disorders that would interfere with cooperation with the requirements of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
VGPR | 4 months
  Very good partial response rate (VGPR) or better after 4 cycles of Dara-CyBorD
Renal Response Rate (RRR) | 4 months
  Renal response rate (RRR, defined as > 30% improvement in creatinine clearance - CrCl from baseline at the point of study entry) after 4 cycles of Dara-CyBorD

SECONDARY OUTCOMES:
Overall response rate (ORR) | 4 months
  Overall response rate (ORR) after 4 cycles of Dara-CyBorD
VGPR, CR, & MRD | 4 months
  Proportion of patients achieving VGPR, CR, and measurable residual disease negativity <10-5 (MRD-), if applicable, after 4 cycles of Dara-CyBorD
Duration of response (DOR) | 2 years
  Duration of response (DOR), defined from the date response achieved to the date of disease relapse
Time to renal response | 2 years
  Time to renal response, defined as the number of days from starting treatment to >30% improvement of CrCl from CrCl at study entry or achieving dialysis independence
Dialysis independence | 4 months
  Proportion of participants who achieved dialysis independence after four cycles of Dara-CyBorD
autologous stem cell transplantation (ASCT) | 4 months
  Proportion of patients undergoing autologous stem cell transplantation (ASCT) after 4 cycles of Dara-CyBorD induction

CONTACTS AND LOCATIONS:
Overall Officials: Amany RA Keruakous, MD, Principal Investigator — Augusta University
Locations (1):
- Georgia Cancer Center-Augusta University, Augusta, Georgia, United States